CLINICAL TRIAL: NCT02788461
Title: A Randomized Phase II Trial to Assess the Efficacy and Safety of Selective Metabolically Adaptive Radiation Dose Escalation in Locally Advanced Non-Small Cell Lung Cancer Receiving Definitive Chemoradiotherapy
Brief Title: Assessing the Efficacy and Safety of Selective Metabolically Adaptive Radiation Dose Escalation in Locally Advanced Non-Small Cell Lung Cancer Receiving Definitive Chemoradiotherapy
Acronym: PET-BOOST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PET-BOOST NSCLC
Record Dates: First submitted 2016-04-28; First posted 2016-06-02 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoradiotherapy (Active Comparator): Patients randomized to the standard arm will receive radiotherapy (5x per week) of 60 gray (Gy) in 30 fractions with concurrent cisplatin and etoposide chemotherapy.
  Interventions: Radiation: Chemoradiotherapy
- Chemoradiotherapy with Integrated Boost Dose (Experimental): Patients randomized to the experimental arm will receive radiotherapy (5x per week) with an integrated boost dose of up to 85Gy in 30 fractions to tumor subvolumes, with concurrent cisplatin and etoposide chemotherapy.
  Interventions: Radiation: Chemoradiotherapy with Integrated Boost Dose

INTERVENTIONS:
Radiation: Chemoradiotherapy — Patients will receive radiotherapy of 60Gy in 30 fractions (5x per week) with concurrent cisplatin and etoposide chemotherapy.
  Arms: Chemoradiotherapy
Radiation: Chemoradiotherapy with Integrated Boost Dose — Patients will receive an RT integrated boost to tumor subvolumes (max boost dose of 85Gy) in 30 fractions (5x per week) with concurrent cisplatin and etoposide chemotherapy.
  Arms: Chemoradiotherapy with Integrated Boost Dose

SUMMARY:
A randomized phase II trial to assess the efficacy and safety of selective metabolically adaptive radiation dose escalation in locally advanced non-small cell lung cancer receiving definitive chemoradiotherapy. Eligible and consenting patients will be randomized to receive conventional chemoradiotherapy or chemoradiotherapy with a radiation (RT) integrated boost. All patients will receive a fludeoxyglucose-positron emission tomography (FDG-PET) scan within two weeks prior to starting treatment. The primary outcome is to determine if dose escalation to metabolically active tumor subvolumes will reduce local-regional failure rate at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years old and are able to consent
* Patients who will undergo Chemo-RT as primarily modality of treatment
* Patients with a primary tumor or node measuring at least 10mm on CT scan
* Patients with a PET avid tumor having Standardized Uptake Values (SUV) > 4
* Patients with Eastern Cooperative Oncology Group (ECOG) status 0-2 within 4 weeks of randomization

Exclusion Criteria:

* Trimodality patients who have surgery as part of curative treatment
* Previous radiotherapy to intended treatment volumes
* Active invasive malignancy other than lung cancer
* Active pregnancy
* Poor respiratory function (Forced Expiratory Volume < 1.0 or Diffusing Capacity < 50% age-adjusted normal)
* ECOG status > 2
* Pre-treatment complete blood count/differential showing inadequate bone marrow reserve (absolute neutrophil count < 1800 cells/mm3 or platelets < 100 000 cells/mm3 or hemoglobin < 90g/L), measured within 4 weeks of registration
* AST, ALT or total bilirubin > 2.5 times the upper limit of normal, measured within 4 weeks of registration
* Unintentional weight loss >10% over 3 months within 4 weeks of registration
* Severe active co-morbidity defined by:
* Significant history of uncontrolled cardiac disease; i.e. uncontrolled hypertension, unstable angina, myocardial infarction within the last 6 months, uncontrolled congestive heart failure, cardiomyopathy with decreased ejection fraction
* Transmural myocardial infection requiring intravenous antibiotics at the time of registration
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before randomization
* Acquired immune deficiency syndrome (AIDS) based on the current Centre for Disease Control definition; note, however, that HIV testing is not required for entry into this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-05; Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Reduction of local-regional failure rate | 2 years
  Primary outcome of the trial is to determine if dose escalation to metabolically active subvolumes will reduce local-regional failure rate

SECONDARY OUTCOMES:
Progression-Free Survival | 2 years
  Determine if dose escalation to metabolically active subvolumes will improve progression-free survival at 2 years
Overall Survival | 2 years
  Determine if dose escalation to metabolically active subvolumes will improve overall survival at 2 years
Grade 3-5 Toxicity Rate | 2 years
  Determine if dose escalation to metabolically active subvolumes will increase the rate of grade 3-5 toxicities
Quality of Life FACT-L | 2 years
  Compare the quality of life in the two arms using Functional Assessment of Cancer Therapy-Lung (FACT-L) instrument
Quality of Life EQ-5D | 2 years
  Compare the quality of life in the two arms using EuroQol Quality of Life-5 Dimensions (EQ-5D) instrument
Dose-Response Characterization | 2 years
  Characterize the tumor dose-response relationship in the experimental arm and create a tumor control probability model for local-regional failure at 2 years
Dose Escalation Feasibility | 2 weeks
  Explore the feasibility of adaptive dose escalation based on PET response at week 2
Imaging Use | 2 years
  Explore the use of Week 0 and Week 2 PET images for prognostication and response assessment for local-regional failure at 2 years

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Cancer Centre at Southlake Regional Health Centre, Newmarket, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Glen site Cedars Cancer Center, Montreal, Quebec
  - CHU de Quebec - L'Hôtel-Dieu de Québec, Québec, Quebec
  - CHUS - Hôpital Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raman S, Bissonnette JP, Warner A, Le L, Bratman S, Leighl N, Bezjak A, Palma D, Schellenberg D, Sun A. Rationale and Protocol for a Canadian Multicenter Phase II Randomized Trial Assessing Selective Metabolically Adaptive Radiation Dose Escalation in Locally Advanced Non-small-cell Lung Cancer (NCT02788461). Clin Lung Cancer. 2018 Sep;19(5):e699-e703. doi: 10.1016/j.cllc.2018.05.002. Epub 2018 May 16. PMID 29903551